CLINICAL TRIAL: NCT02774954
Title: Preventing Injection Initiation: The Change the Cycle Randomized Controlled Trial.
Brief Title: Change the Cycle: An RCT to Prevent Injection Initiation
Acronym: CTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); RTI International (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Ricky Bluthenthal, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-15-00243; R01DA038965 (NIH)
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Substance Abuse, Intravenous; HIV; Heroin Dependence; Opioid Dependence; Cocaine Dependence; Amphetamine Dependence
Keywords: Change the cycle; social learning theory; people who inject drugs; injection drug use; Information, Motivation, Behavior Skills Model; Longitudinal cohort study
MeSH Terms: conditions — Substance Abuse, Intravenous; Heroin Dependence; Opioid-Related Disorders; Cocaine-Related Disorders; Amphetamine-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study compares 2 active listening, information-motivation-behavior skills interventions aimed at improving health behaviors among very low-income, drug using participants.
Who Masked: Outcomes Assessor
Masking Description: The statistician who is conducting the data analysis will not know the content of the intervention assignment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Change the cycle (Experimental): CTC uses the Information-Motivation-Behavioral skills (IMB) model to achieve changes among active PWID through seven short modules. Information and motivational domains are addressed in guided conversations about (1) their own first injection episode and consequences, (2) past experiences initiating injection-naive people and consequences, (3) health, legal, and social risks related to injection drugs, (4) health, legal, social risks of initiating people, and (5) identifying their own behaviors that might promote injection among others. The behavioral skills domain is addressed through a (6) skill-building discussion and rehearsal of responses to possible initiation scenarios, and (7) safer injection education.
  Interventions: Behavioral: Change the Cycle
- Nutrition (Active Comparator): The nutrition equal attention control intervention is a single-session, 60- minute Information-Motivation-Behavioral (IMB) skills-based intervention addressing healthy eating. The healthy eating intervention uses a one-on-one guided conversation between the interventionist and the participant. The intervention addresses (1) information about current eating patterns and recommendations for healthy alternatives (20 minutes), (2) motivations for improving healthy eating by providing feedback to participants on personal responsibility, a menu of alternative change options, a decision balance exercise, and eating goal setting (10 minutes), and (3) Behavioral Self-Management Component (30 minutes) that covers eating scenarios, participant responses, and healthy alternatives to the scenario and the participants feedback.
  Interventions: Behavioral: Change the Cycle

INTERVENTIONS:
Behavioral: Change the Cycle — See previous response
  Other Names: CTC

SUMMARY:
The study will test the efficacy of a hour long, one-on-one, active listening counseling session (called Change the Cycle or CTC) aimed at reducing behaviors among active people who inject drugs (PWID) that research has found to facilitate uptake of injection drug use among non-injectors. The study will involve ~1,100 PWID who will be randomized to CTC or an equal attention control intervention on improving nutrition. Participants will be recruited in Los Angeles and San Francisco, California and followed up at 6 and 12 months to determine changes in direct and indirect facilitation of injection initiation among non-injectors.

DETAILED DESCRIPTION:
The study goal is to conduct a large-scale randomized controlled trial (RCT) of the "Change the Cycle" (CTC) intervention. CTC is an hour long, single-session, one-on-one intervention that aims to reduce injection initiation by encouraging active PWID to not promote drug injection, model injection behavior, describe how to inject, or assist in injection initiations of non-injectors. CTC uses the Information-Motivation-Behavioral skills (IMB) model to achieve changes among active PWID through seven short modules. Information and motivational domains are addressed in guided conversations about (1) their own first injection episode and consequences, (2) past experiences initiating injection-naive people and consequences, (3) health, legal, and social risks related to injection drugs, (4) health, legal, social risks of initiating people, and (5) identifying their own behaviors that might promote injection among others. The behavioral skills are addressed through (6) skill-building discussions and consideration of common initiation scenarios, and (7) safer injection education.

Aim 1: To test the efficacy of CTC on reducing the number of non-injectors initiated into injection (counts) by PWID. Hypothesis 1: PWID who receive CTC will report initiating fewer non-injectors into drug injection at 6 and 12 months as compared with PWID in the control condition.

Aim 2: To test the efficacy of CTC on reducing the number of times PWID are asked to initiate (counts) someone into injection. Hypothesis 2: PWID who receive CTC will report having been asked fewer times to initiate someone into drug injection at 6 and 12 months as compared with PWID in the control condition.

Aim 3: To test whether injection initiation social learning risks (injecting in front of, describing injection to, and speaking positively about injection to non-injectors) act as mediational mechanisms for the efficacy of the CTC intervention on initiation and request-to-initiate outcomes. Hypothesis 3: Social learning variables will significantly mediate the association between the CTC intervention and episodes of initiating and being requested to initiate someone into drug injection at 6 and 12 months.

To achieve these aims, active PWID (N=1,076) will be randomly assigned to receive CTC or an equal attention control condition in Los Angeles (LA) and San Francisco (SF), CA. Injection initiation and injection initiation social learning variables will be collected at baseline, 6 months, and 12 months using computer-assisted personal-interviewing (CAPI). The equal attention control condition will focus on improving nutrition, specifically increasing fresh water intake and protein consumption, and will replicate CTC in length, theoretical foundation (IMB), and modality (1 on 1 personal session).

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Injection an illicit drug in the last 30 days,
* visible evidence of injection such as track mark or stigmata,
* at least 18 years of age

Exclusion Criteria:

* Under 18 years of age,
* no self-reported drug injection in the last 30 days,
* no physical evidence of recent drug injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 979 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricky Bluthenthal, PhD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - RTI International, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
Using the National Addiction and HIV Data Archive program (NAHDAP), we will provide our datasets and codebooks to researchers in a format that facilitates data-sharing. After the completion of the study, the dataset will be de-identified and made available for secondary analysis on the NAHDAP website (http://www.icpsr.umich.edu/icpsrweb/NAHDAP/). Researchers who request access will be given a password to access the data, documentation, and surveys. As part of the registration process, researchers will sign an agreement to adhere to the data coding guidelines that were developed for the project, will state their intentions for use, and will agree to inform the original investigators of their findings and publications for tracking purposes with acknowledgments to the granting agency. Because the respondents will be identified only by ID codes in the datasets, it will be impossible to identify individuals from the datasets.
Supporting Information: Study Protocol, ICF
Time Frame: June 2020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in community settings using targeted sampling approach. The first participant was recruited on June 20, 2016 and the last participant was recruited on October 1, 2017.
Pre-assignment Details: A total of 984 participants were recruited of whom 979 complete baseline study requirements and are considered in the trial.
Period: Baseline
Arm/Group | Change the Cycle | Nutrition
Started | 482 | 497
Completed Baseline Interview and Intervention | 482 | 497
Completed | 482 | 497
Not Completed | 0 | 0
Period: 6 Month Follow-up
Arm/Group | Change the Cycle | Nutrition
Started | 482 | 497
Completed | 286 | 313
Not Completed | 196 | 184
Period: 12 Month Follow-up
Arm/Group | Change the Cycle | Nutrition
Started | 286 | 313
Completed | 253 | 279
Not Completed | 33 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Change the Cycle | Nutrition | Total
Number analyzed (Participants) | 482 | 497 | 979
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 467 | 484 | 951
  >=65 years | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.44 (12.22) | 42.17 (12.12) | 42.30 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 118 | 223
  Male | 377 | 379 | 756
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 125 | 120 | 245
  Not Hispanic or Latino | 357 | 377 | 734
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 28 | 33 | 61
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 94 | 106 | 200
  White | 332 | 326 | 658
  More than one race | 22 | 27 | 49
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 482 | 497 | 979
People helped inject for the first time in the last 6 months [Mean (Standard Deviation); unit: Number of people] | 5.14 (13.65) | 6.72 (25.00) | 5.94 (20.13)
Number of people who asked to be initiated in the last 6 months [Mean (Standard Deviation); unit: Number of people] | 11.09 (13.65) | 10.45 (41.50) | 10.77 (36.93)

OUTCOME MEASURES:

1. Primary Outcome: People Initiated Into Injection Drug Use
Description: This data is collected based on responses to the following question: "In the last 6 months, how many people have you helped injected for the first time?"
Time Frame: 6 months
Population: Participants in the study are people who inject drugs.
Measure: Mean (Standard Deviation); unit: People initiated
Arm/Group | Change the Cycle | Nutrition
Number analyzed (Participants) | 253 | 279
People initiated | 2.05 (1.43) | 3.26 (5.43)
Statistical Analysis 1: Comparison: Change the Cycle; Test type: Superiority; p = 0.35, ANOVA

2. Primary Outcome: Number of Request to Initiate Someone Into Drug Injection
Description: This data is collected based on responses to the following question: "In the last 6 months, has anyone ASKED you to help them inject an illicit drug for the first time?"
Time Frame: 6 months
Population: Participants are people who inject drugs. The outcomes variable is the number of people who requested that participants help them with their first injection drug use. Study participants could receive multiple request.
Measure: Mean (Standard Deviation); unit: Initiation request
Arm/Group | Change the Cycle | Nutrition
Number analyzed (Participants) | 253 | 279
Initiation request | 6.42 (25.48) | 4.06 (5.56)
Statistical Analysis 1: Comparison: Change the Cycle; Test type: Superiority; p = 0.35, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were tracked for the participants time in the study which could have extended up to 18 months.
Arm/Group | Change the Cycle | Nutrition
All-Cause Mortality (participants affected / at risk) | 17/482 | 17/497
Serious Adverse Events (participants affected / at risk) | 0/482 | 0/497
Other Adverse Events (participants affected / at risk) | 0/482 | 0/497

LIMITATIONS AND CAVEATS:
Our chief limitation was loss-to-follow-up. Our rate of recapture at 6 month was 62% while are recapture rate between 6 month and 12 month interview was 89%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT02774954/Prot_SAP_000.pdf